CLINICAL TRIAL: NCT05128266
Title: Broken Endodontic Instrument Removal Using Ultrasounds, Microscope and a Modified Spinal Needle
Brief Title: Broken Instrument Removal
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Carlo Lajolo, Associate Professor and Principal Investigator, Catholic University of the Sacred Heart
Other Study IDs: Oss-R-233
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Endodontically Treated Teeth; Endodontical Retreatment
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endodontical Retreatment: non-surgical retreatment of teeth with broken file instrument into the canal using ultrasounds, microscope and a modified spinal needle
  Interventions: Procedure: Endodontical Retreatment

INTERVENTIONS:
Procedure: Endodontical Retreatment — 1. Linear canal Removal of the coronal dentine in order to create the space useful to an extractor to catch and remove the instrument. The preferred instrument to reach this aim is a .15 or .20 ultrasonic tip.
  2. Curve canal When the instrument is broken inside a curve canal, it is not possible to create a circumferential space around the separated instrument without the risk of root perforation. Thus, the first step is the removal of the dentine of the external wall of the root canal. The second step is the removal of the dentine of the internal wall of the root canal. This selective removal of dentinal tissue unlocks thee separated instrument and determines its mobilization. Thus, the irrigation itself makes the instrument available for the removal.
  After the removal of the broken instrument, root canal preparation was completed Canal filling was performed based on Schilder's technique.

SUMMARY:
The aims of this retrospective analysis are (1) to evaluate the success rate of a non-surgical retreatment of teeth with broken file instrument into the canal using ultrasounds, microscope and a modified spinal needle, (2) to assess the outcome of the treatment if the remaining fragment was left, bypassed or removed from the root canal in terms of survival rate of the treated teeth after a 5-years follow up period.

DETAILED DESCRIPTION:
The fracture of an endodontic instrument is a frustrating phenomenon, both for practitioners and patients, that can compromise the cleaning and shaping procedures of the root canal treatment, with a potential impact on the treatment outcome. In the past decades, the advent of rotary nickel titanium instruments resulted in an increased incidence of instrument separation.

Two mechanisms have been reported in order to describe the fracture of an endodontic instrument inside the root canal: torsional stress and cyclic fatigue. Cyclic failure is due to the constant tension and compression which insists on the file when it shapes the maximal root canal curvature area. Torsional failure occurs when the tip of the instrument locks on the wall of the root canal while the shafts keeps rotating, and the torque exceeds the plastic limit of the metal.

Several studies focused on causes and factors influencing the weakening of endodontic instrument after clinical use, and some recommendation were given trying to minimized the risk of instruments breakage. Nevertheless, this problem can still occur, even to an experienced operator, making the achievement of a correct and predictable root canal final treatment uncertain.

Due to their complexity, many of these cases are approached by extraction and implant replacement of the so evaluated "hopeless" tooth. Treatment decisions can vary widely among dentists and dental specialists and may be based more on personal values and experience than an objective analysis of treatment benefits, risks, costs, prognosis, and alternatives.

At present, there is no standardized procedure for safe and consistently successful instrument fragment removal in the dental literature.

Different devices, techniques, methods, and protocols used for removal of separated instruments are described in literature. Unfortunately, there is a lack of high-level evidence, since most of the papers refer to clinical case report.

Until the beginning of endodontics, dentists have had to face this problem and already in the last century Masserann invented an instrument to remove obstacles in the root canals. Some authors believe that Masserann instrument used by expert hands does not expose the tooth to the root fracture, but this risk remains very high. Several other instruments were invented as a result, many of them similar to the Masserann extractor, others using micro tweezers or cyanoacrylate glue.

To solve the problem of root canal obstruction due to fragments of root canal instruments, some authors make use of the technique of intentional reimplantation after retreatment of the tooth out of the mouth. Recently, some authors have also used the Nd: YAG laser to remove broken instruments in the canals. Laser energy has been used to melt the solder, connecting the separated instrument with the brass tube.

Furthermore, the literature is not clear about the actual need to remove the instruments from the root canals, neither about the percentage of successes in case of bypassing the fragment or about the persistence of the instrument in the root canal.

Independently from the technique, the optimal management of instrument fragments during root canal treatment is crucial in order to enable sufficient debridement and obturation of the root canal system. However, all clinicians agree that the best help in this procedure came by the combined use of ultrasound and the operative microscope. These two devices used in combination allow a more efficient and accurate work, lowering the risk of weakening the canal wall or create root perforations.

The aims of this retrospective analysis are (1) to evaluate the success rate of a non-surgical retreatment of teeth with broken file instrument into the canal using ultrasounds, microscope and a modified spinal needle, (2) to assess the outcome of the treatment if the remaining fragment was left, bypassed or removed from the root canal in terms of survival rate of the treated teeth after a 5-years follow up period.

ELIGIBILITY:
Inclusion Criteria:

All patients who received an endodontic retreatment due to a separated instrument inside a root canal were included in this study.

Exclusion Criteria:

Exclusion criteria were unavailability of complete clinical data or the use of other retreatment techniques.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients needing an endodontic retreatment due to a separated instrument inside a root canal.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 1991-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Success rate of a non-surgical retreatment | after 5-years follow-up
  Number of non extracted teeth

SECONDARY OUTCOMES:
Influence of the type of Tooth on the outcome of the treatment | After 5-years follow-up
  Molar, Premolar, Canine, Incisor
Influence of the type of Root Canal on the outcome of the treatment | After 5-years follow-up
  Curve or Linear Canal
Influence of the corono-apical level of the fracture on the outcome of the treatment | After 5-years follow-up
  Coronal, Medium, Apical third of the root canal
Influence of the presence of periapical lesion on the outcome of the treatment | After 5-years follow-up
  Yes or Not
Influence of the presence of a root fracture on the outcome of the treatment | After 5-years follow-up
  Yes or Not
Influence of the presence of a root perforation on the outcome of the treatment | After 5-years follow-up
  Yes or Not

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Malentacca A, Zaccheo F, Rupe C, Lajolo C. Endodontic Clinical Outcome after Separated Instrument Removal Using a Spinal Needle Technique: A Retrospective Study of Thirty Years of Clinical Experience. J Endod. 2023 Aug;49(8):980-989. doi: 10.1016/j.joen.2023.06.007. Epub 2023 Jul 7. PMID 37422250